CLINICAL TRIAL: NCT03452644
Title: Diagnostic Yield of Ultrasound-Guided Needle Biopsy in the Diagnosis of Musculoskeletal Soft-Tissue Tumors
Brief Title: US-Guided Biopsy in the Diagnosis of Musculoskeletal Soft-Tissue Tumors
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Alberto Bazzocchi, Dr., Istituto Ortopedico Rizzoli
Other Study IDs: Softbiopsy@IOReco
Record Dates: First submitted 2018-02-23; First posted 2018-03-02 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Soft Tissue Neoplasm; Soft Tissue Sarcoma; Soft Tissue Mass; Soft Tissue Lesion
Keywords: US-CNB; Soft Tissue Mass; Soft Tissue Sarcoma; Soft Tissue Neoplasm; Soft Tissue Lesion
MeSH Terms: conditions — Soft Tissue Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective evaluation of soft tissue tumors that have undergone core needle biopsy with US guidance (US-CNB)

DETAILED DESCRIPTION:
The present study is designed to be the first step in the creation of an interdisciplinary platform collecting data on patients and procedures to provide a predictive tool to help physicians in the management of patients affected by a soft tissue lesion.

The primary aim of our work is to evaluate the diagnostic yield of US-CNB. The secondary aim is to exploit all the imaging data conventionally available at a Sarcoma Center before a biopsy on a soft tissue mass, to build a multiparametric model and score of prediction of malignancy, and eventually of biological behavior - grading.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone US-CNB for soft tissue lesions at the Rizzoli Orthopaedic Institute

Exclusion Criteria:

* Patients whose histological diagnosis is not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll 350 patients who underwent US-CNB for soft tissue lesion at the Rizzoli Orthopaedic Institute
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | One year
  Diagnostic yield will be defined as the number of diagnostic core needle biopsies divided by the total number of core needle biopsies. A diagnostic yield > 94% will be considered sufficient to produce a sample to reach the histological diagnosis.

SECONDARY OUTCOMES:
Prediction of malignancy | One year
  To determine which imaging features and biomarkers correlates with malignancy and biological behavior of soft tissue masses.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Bazzocchi, MD, PhD, Principal Investigator — The Rizzoli Ortopaedic Institute
Locations (1):
- The Rizzoli Orthopaedic Institute, Bologna, Bo, Italy

IPD SHARING:
Plan to Share IPD: No